CLINICAL TRIAL: NCT04052347
Title: Decision Aid to Assist Low-Risk Nulliparous Women Considering Induction of Labor At 39 Weeks: A Randomized Trial (DAWN Trial)
Brief Title: Decision Aid to Assist Low-Risk Nulliparous Women Considering Induction of Labor At 39 Weeks
Acronym: DAWN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid related
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sunbola S Ashimi Ademola, Senior Researcher, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-19-0490
Record Dates: First submitted 2019-07-15; First posted 2019-08-09 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Pregnancy Related; Elective Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared decision-making with a patient decision-aid (Experimental)
  Interventions: Behavioral: Shared decision-making with a Decision-aid
- routine shared decision-making (Active Comparator): control group
  Interventions: Behavioral: routine shared decision-making

INTERVENTIONS:
Behavioral: Shared decision-making with a Decision-aid — A tablet computer-based decision-aid was developed by the study investigators based on the standards of the International Patient Decision Aid Standards Collaboration9
  Arms: Shared decision-making with a patient decision-aid
Behavioral: routine shared decision-making — control group
  Arms: routine shared decision-making

SUMMARY:
The primary objective is to assess if the utilization of a decision-aid increases the likelihood of low-risk nulliparous women undergoing elective induction of labor at 39.0-39.6 weeks

ELIGIBILITY:
Inclusion Criteria:

* Low-risk nulliparous women- no previous pregnancy > 23 weeks
* 18-50 years of age
* Singleton gestation
* Between 34.0 and 36.6 weeks at the time of screening. Randomization must occur between 37.0-37.6 weeks inclusive.

Exclusion Criteria:

* 1. First sonographic examination after 20 weeks 2. Women with any of the following comorbidities (at the time of randomization):

  1. Autoimmune disorders (antiphospholipid antibody, lupus, rheumatoid arthritis, scleroderma)
  2. Cerclage in the index pregnancy
  3. Diabetes mellitus-gestational or pre-gestational
  4. Hematologic disorders (coagulation defects, sickle cell disease, thrombocytopenia, thrombophilia)
  5. Hypertension (chronic or pregnancy induced) before enrollment
  6. HIV (human immunodeficiency virus)
  7. Institutionalized individuals (prisoners)
  8. Prior obstetric history of: 1) intrauterine growth restriction, 2) preterm birth before 34 weeks, 3) severe preeclampsia, eclampsia, HELLP syndrome, and 4) stillbirth after 24 weeks or neonatal death
  9. Preterm labor or ruptured membranes before enrollment
  10. Psychiatric disorder (bipolar, depression) on medication
  11. Placenta previa / 3rd trimester bleeding
  12. Renal insufficiency (serum creatinine > 1.5 mg/dL)
  13. Restrictive lung disease
  14. Fetal red blood cell isoimmunization
  15. Seizure disorder on medication
  16. Thyroid disease on medication
  17. Body Mass Index (BMI) above 40 kg/m 3. Major fetal Anomaly including: anencephaly, spina bifida, bilateral renal agenesis, cystic hygroma with hydrops, diaphragmatic hernia, or congenital heart defects 4. Unable to understand consent in English or Spanish

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects who decided to undergo elective induction of labor at 39.0-39.6 weeks after utilization of a decision-aid | 4 weeks
  Number of subjects who decided to undergo elective induction of labor at 39.0-39.6 weeks after utilization of a decision-aid

SECONDARY OUTCOMES:
Composite neonatal morbidity | at delivery
  Composite neonatal morbidity among (CNM) is any of the following: 1) Apgar score < 7 at 5 min, 2) umbilical arterial pH < 7.00, 3) intraventricular hemorrhage grade III or IV, 4) periventricular leukomalacia, 5) intubation for over 24 hrs, 6) necrotizing enterocolitis grade 2 or 3, 7) stillbirth or 8) death within 28 days of birth.
Maternal morbidities | 1 week
  Number of subjects with morbidities as described by American College of Obstetrics and Gynecology (ACOG)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No